CLINICAL TRIAL: NCT01978717
Title: General Anesthesia Combined With Epidural Anesthesia Mitigates the Surgical Stress-related Immunosuppression in Patients With Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhong Miao (Other)
Responsible Party: Sponsor-Investigator, Changhong Miao, Professor, Department of Anesthesiology, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO.2011-197; 08431910200 (Other Grant/Funding Number: Shanghai Municipal Science and Technology Commission)
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Colorectal Neoplasms
Keywords: Anesthesia; T-helper; MDSCs; Colorectal cancer; Fast track
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Anesthesia, Epidural; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- general anesthesia & epidural anesthesia (Experimental): 26 patients received general anesthesia combined with epidural anesthesia for surgery, and patient-controlled epidural analgesia for 2 days after surgery
  Interventions: Procedure: epidural anesthesia; Procedure: general anesthesia
- general anesthesia (Experimental): 27 patients received general anesthesia for surgery, and patient-controlled intravenous analgesia for 2 days after surgery
  Interventions: Procedure: general anesthesia

INTERVENTIONS:
Procedure: epidural anesthesia
  Arms: general anesthesia & epidural anesthesia
Procedure: general anesthesia — Patients received general anesthesia for surgery

SUMMARY:
The purpose of this study is to prove whether general anesthesia combined with epidural anesthesia could better maintain body balance of Th1/Th2 and Treg/Th17 compared with general anesthesia, so as to reduce the surgical stress-related immunosuppression, and to improve the prognosis.

ELIGIBILITY:
Inclusion Criteria:

* patients with Colorectal Cancer(CRC);
* subjected to the Fast-Track processing of surgery;
* between 18 and 75 years old.

Exclusion Criteria:

* American Society of Anesthesiologists(ASA) grade > III;
* BMI > 30;
* a history of abdominal surgery, endocrine or immune system dysfunction;
* recent blood transfusions, hormone or non-steroidal anti-inflammatory therapy during the past month;
* previous contraindication to epidural anesthesia.

Ages: 51 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The changes of peripheral immune cells and cytokines | within the first 5 days after surgery
  The changes of peripheral subtype of T-helper, myeloid-derived suppressor cells(MDSCs) and cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- Zhong Shan Hospital Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Chen WK, Miao CH. The effect of anesthetic technique on survival in human cancers: a meta-analysis of retrospective and prospective studies. PLoS One. 2013;8(2):e56540. doi: 10.1371/journal.pone.0056540. Epub 2013 Feb 20. PMID 23437162